CLINICAL TRIAL: NCT02253251
Title: Clinical Validation of the Role of microRNA Binding Site Mutations in Cancer Risk, Prevention and Treatment
Status: Recruiting | Type: Observational
Sponsor: MiraKind (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00009633
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cancer
Keywords: Breast Cancer; Cancer Risk; Family Breast and Ovarian Cancer; Genetic Cancer Risk; Cancer Treatment; Familial multiple primary cancer risk; Autoimmunity; Endometriosis
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Autoimmune Diseases; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — DNA will be isolated from the submitted sample and kept with permission for additional studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Family Registry: For individuals identified with the KRAS-variant. Patients will be prospectively followed to determine the impact of lifestyle on disease risk.
  Interventions: Genetic: KRAS-variant and microRNA binding site mutation testing
- Double primary breast cancer: Women with multiple primary breast cancer will be tested for the KRAS-variant and compared between those with this mutation and those without.
  Interventions: Genetic: KRAS-variant and microRNA binding site mutation testing
- Autoimmunity: We have shown that the KRAS-variant and other members of this genetic class of mutations associate with altered immunity, leading to immunosuppression as well as autoimmunity.
  Interventions: Genetic: KRAS-variant and microRNA binding site mutation testing
- Cancer patients receiving certain treatments: We have found that microRNA binding site mutations are predictive biomarkers of outcomes from cancer therapy, including response and toxicity. We will enroll patients to further study and validate these findings.
  Interventions: Genetic: KRAS-variant and microRNA binding site mutation testing

INTERVENTIONS:
Genetic: KRAS-variant and microRNA binding site mutation testing — Participant in these studies will be tested for the KRAS-variant

SUMMARY:
The investigators will recruit and enroll individuals that may have the KRAS-variant or other microRNA binding site mutations to join registry studies. The investigators will allow individuals to obtain their results through a physician at the completion of the studies. The investigators current focus is cancer and autoimmunity.

DETAILED DESCRIPTION:
The investigators have identified germ-line microRNA binding site mutations that predict an increased risk of cancer, endometriosis and associated infertility, and unique tumor biology and response to treatment. The goal of this protocol is to further determine the mechanisms of these mutations, such as the KRAS-variant, and their associations with human health, such as cancer. The investigators will collect saliva samples from individual patients who are eligible and choose to enroll in these studies, to test for the KRAS-variant and/or other mutations under study. With specific permission, the investigators will keep excess DNA to further investigate and discover additional similar mutations. The investigators purpose is to have participants answer questionnaires about lifestyle factors in an ongoing manner, to understand the impact of different factors on cancer risk for patients with these mutations.

ELIGIBILITY:
Inclusion Criteria:

* Personal or family history of cancer
* Personal history of endometriosis, or autoimmunity

Exclusion Criteria:

* Younger than 18
* Non-english speaking and unable to understand and sign the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast and ovarian cancer patients and the family members of those that have the KRAS-variant from primarily the US. Those with Autoimmunity.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2014-09; Primary Completion 2030-12 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Measuring the prevalence of the KRAS-variant in certain populations Prevalence of the KRAS-variant in BRCA negative breast cancer patients | 1 year
  The Prevalence of the KRAS-variant will be determined in specific populations, such as women with drug resistant endometriosis, or BRCA negative breast cancer. The prevalence will be compared to extensive data on the expected and known prevalence of the KRAS-variant in non-diseased populations. Statistical significance will be determined by Chi-squared analysis.
Comparing the impact of interventions in KRAS-variant versus non-KRAS variant populations | 1 year
  We will compare the impact of specific treatment approaches for example in women with the KRAS-variant and double primary breast cancer, versus the interventions used in non-KRAS-variant double primary breast cancer patients.

SECONDARY OUTCOMES:
The impact of lifestyle factors on cancer risk for KRAS-variant patients | 10 years
  Individuals with the KRAS-variant will be prospectively followed, and lifestyle factors will be associated with changes in health, including cancer development. Our goal is to compare baseline characteristics between individuals with the KRAS-variant who do, versus do not, develop cancer, for example.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Weidhaas, MDPhD, Principal Investigator — MiraKind
Locations (1):
- MiraKind, Los Angeles, California, United States

REFERENCES:
- [Background] Saridaki Z, Weidhaas JB, Lenz HJ, Laurent-Puig P, Jacobs B, De Schutter J, De Roock W, Salzman DW, Zhang W, Yang D, Pilati C, Bouche O, Piessevaux H, Tejpar S. A let-7 microRNA-binding site polymorphism in KRAS predicts improved outcome in patients with metastatic colorectal cancer treated with salvage cetuximab/panitumumab monotherapy. Clin Cancer Res. 2014 Sep 1;20(17):4499-4510. doi: 10.1158/1078-0432.CCR-14-0348. PMID 25183481
- [Background] Chung CH, Lee JW, Slebos RJ, Howard JD, Perez J, Kang H, Fertig EJ, Considine M, Gilbert J, Murphy BA, Nallur S, Paranjape T, Jordan RC, Garcia J, Burtness B, Forastiere AA, Weidhaas JB. A 3'-UTR KRAS-variant is associated with cisplatin resistance in patients with recurrent and/or metastatic head and neck squamous cell carcinoma. Ann Oncol. 2014 Nov;25(11):2230-2236. doi: 10.1093/annonc/mdu367. Epub 2014 Jul 31. PMID 25081901
- [Background] Pilarski R, Patel DA, Weitzel J, McVeigh T, Dorairaj JJ, Heneghan HM, Miller N, Weidhaas JB, Kerin MJ, McKenna M, Wu X, Hildebrandt M, Zelterman D, Sand S, Shulman LP. The KRAS-variant is associated with risk of developing double primary breast and ovarian cancer. PLoS One. 2012;7(5):e37891. doi: 10.1371/journal.pone.0037891. Epub 2012 May 25. PMID 22662244
- [Background] Grechukhina O, Petracco R, Popkhadze S, Massasa E, Paranjape T, Chan E, Flores I, Weidhaas JB, Taylor HS. A polymorphism in a let-7 microRNA binding site of KRAS in women with endometriosis. EMBO Mol Med. 2012 Mar;4(3):206-17. doi: 10.1002/emmm.201100200. Epub 2012 Feb 3. PMID 22307873
- [Background] Ratner ES, Keane FK, Lindner R, Tassi RA, Paranjape T, Glasgow M, Nallur S, Deng Y, Lu L, Steele L, Sand S, Muller RU, Bignotti E, Bellone S, Boeke M, Yao X, Pecorelli S, Ravaggi A, Katsaros D, Zelterman D, Cristea MC, Yu H, Rutherford TJ, Weitzel JN, Neuhausen SL, Schwartz PE, Slack FJ, Santin AD, Weidhaas JB. A KRAS variant is a biomarker of poor outcome, platinum chemotherapy resistance and a potential target for therapy in ovarian cancer. Oncogene. 2012 Oct 18;31(42):4559-66. doi: 10.1038/onc.2011.539. Epub 2011 Dec 5. PMID 22139083
- [Background] Lee LJ, Ratner E, Uduman M, Winter K, Boeke M, Greven KM, King S, Burke TW, Underhill K, Kim H, Boulware RJ, Yu H, Parkash V, Lu L, Gaffney D, Dicker AP, Weidhaas J. The KRAS-variant and miRNA expression in RTOG endometrial cancer clinical trials 9708 and 9905. PLoS One. 2014 Apr 14;9(4):e94167. doi: 10.1371/journal.pone.0094167. eCollection 2014. PMID 24732316
- [Background] Smits KM, Paranjape T, Nallur S, Wouters KA, Weijenberg MP, Schouten LJ, van den Brandt PA, Bosman FT, Weidhaas JB, van Engeland M. A let-7 microRNA SNP in the KRAS 3'UTR is prognostic in early-stage colorectal cancer. Clin Cancer Res. 2011 Dec 15;17(24):7723-31. doi: 10.1158/1078-0432.CCR-11-0990. Epub 2011 Oct 12. PMID 21994416
- [Background] Paranjape T, Heneghan H, Lindner R, Keane FK, Hoffman A, Hollestelle A, Dorairaj J, Geyda K, Pelletier C, Nallur S, Martens JW, Hooning MJ, Kerin M, Zelterman D, Zhu Y, Tuck D, Harris L, Miller N, Slack F, Weidhaas J. A 3'-untranslated region KRAS variant and triple-negative breast cancer: a case-control and genetic analysis. Lancet Oncol. 2011 Apr;12(4):377-86. doi: 10.1016/S1470-2045(11)70044-4. Epub 2011 Mar 22. PMID 21435948
- [Background] Hollestelle A, Pelletier C, Hooning M, Crepin E, Schutte M, Look M, Collee JM, Nieuwlaat A, Dorssers LC, Seynaeve C, Aulchenko YS, Martens JW, van den Ouweland AM, Weidhaas JB. Prevalence of the variant allele rs61764370 T>G in the 3'UTR of KRAS among Dutch BRCA1, BRCA2 and non-BRCA1/BRCA2 breast cancer families. Breast Cancer Res Treat. 2011 Jul;128(1):79-84. doi: 10.1007/s10549-010-1080-z. Epub 2010 Jul 30. PMID 20676756
- [Background] Ratner E, Lu L, Boeke M, Barnett R, Nallur S, Chin LJ, Pelletier C, Blitzblau R, Tassi R, Paranjape T, Hui P, Godwin AK, Yu H, Risch H, Rutherford T, Schwartz P, Santin A, Matloff E, Zelterman D, Slack FJ, Weidhaas JB. A KRAS-variant in ovarian cancer acts as a genetic marker of cancer risk. Cancer Res. 2010 Aug 15;70(16):6509-15. doi: 10.1158/0008-5472.CAN-10-0689. Epub 2010 Jul 20. PMID 20647319
- [Background] Chin LJ, Ratner E, Leng S, Zhai R, Nallur S, Babar I, Muller RU, Straka E, Su L, Burki EA, Crowell RE, Patel R, Kulkarni T, Homer R, Zelterman D, Kidd KK, Zhu Y, Christiani DC, Belinsky SA, Slack FJ, Weidhaas JB. A SNP in a let-7 microRNA complementary site in the KRAS 3' untranslated region increases non-small cell lung cancer risk. Cancer Res. 2008 Oct 15;68(20):8535-40. doi: 10.1158/0008-5472.CAN-08-2129. PMID 18922928
- See also: non-profit running the study — http://mirakind.org